CLINICAL TRIAL: NCT00997750
Title: Prospective Randomized Double-center Study of Nonsteroidal Antinflammatory Drug Lornoxicam in Patients With Acute Coronary Syndrome Without Persistent ST- Segment Elevation
Brief Title: Efficacy and Safety of Lornoxicam in Patients With Acute Coronary Syndrome
Acronym: PLEA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Clinical Hospital w/Outpatient Health Center of Business Administration for the President of Russian Federation (Other Government)
Responsible Party: Dr Nikita Lomakin, Central Clinical Hospital of President Department of Russian Federation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AB-CCH-51
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2009-10-19 (Estimated); Status verified 2009-10

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS; Acute Coronary Syndrome; NSAID; Lornoxicam; Xefocam
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — lornoxicam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lornoxicam (Experimental): Lornoxicam 8mg/day and 12mg/day for 15 days
  Interventions: Drug: Lornoxicam

INTERVENTIONS:
Drug: Lornoxicam — lornoxicam 8mg/day and 12mg/day for 15 days
  Other Names: Xefocam

SUMMARY:
The purpose of this study is to determine whether nonsteroidal antiinflammatory drug lornoxicam in combination with low dose aspirin (100mg/day) is effective and safe in patients with Acute Coronary Syndrome without persistent ST-segment elevation.

DETAILED DESCRIPTION:
Nonsteroidal Antiinflammatory drugs (NSAIDs) are the most frequently prescribed drugs in the world. There are a lot of controversial information published during recent years about NSAID cardiosafety. It is still unclear do NSAIDs develop cardioprotective or cardiotoxic effects in acute and chronic heart disease patients. Aim of the study was to investigate safety and efficacy of Lornoxicam, nonselective COX-inhibitor, in patients with acute coronary syndrome without ST-segment elevation (NSTEACS) and to evaluate the influence of Lornoxicam on C-reactive protein (CRP) and IL-6, IL-10 levels.

ELIGIBILITY:
Inclusion Criteria:

1. Unstable angina verified during first 48 hours after admitting to the hospital or
2. Acute Miocardial infarction without St-segment elevation verified during first 48 hours after admitting to the hospital

Exclusion Criteria:

1. High risk of bleeding of any location
2. Any kind of acute and active inflammatory process (excluding acute coronary syndrome)
3. Aspirin or NSAID Intolerability
4. No informed consent
5. Acute peptic stomach or duodenum ulcer
6. Acute or chronic renal failure (serum creatinin >300 mmol/l)
7. Acute cerebrovascular bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
All Cardiovascular events (cardiovascular dearth+nonfatal miocardial infarction+unstable angina) | six months

SECONDARY OUTCOMES:
Noncardiovascular death, Gastrointestinal bleeding | six months

CONTACTS AND LOCATIONS:
Overall Officials: Alexei K Gruzdev, Prof, Study Chair — Department of Cardiology, Central Clinical Hospital of Presidential Administration of Russian Federation
Locations (1):
- Central Clinical Hospital of Presidential Department Of Russian Federation, Moscow, Russia

REFERENCES:
- [Background] Lomakin N.V., Gruzdev A.K. Cardiovascular risks of cyclooxygenase inhibitors (data review). Kardiol serdecno-sosud hir #1:28-36, 2009 (http://www.mediasphera.ru/journals/cardsurg/530/eng/8095/)